CLINICAL TRIAL: NCT04097548
Title: Psychosocial Intervention, Maternal Inflammation, and Birth Outcomes: Centering vs. Routine Prenatal Care
Brief Title: A RCT of CenteringPregnancy on Birth Outcomes and Maternal Inflammation
Acronym: PIINC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Endeavor Health (Other)
Collaborators: Prisma Health-Upstate (Other); Northwestern University (Other); University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Ann Borders, Principal Investigator, Endeavor Health
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: EH17-256
Record Dates: First submitted 2019-06-26; First posted 2019-09-20 (Actual); Last update posted 2023-11-09 (Actual); Status verified 2023-11

CONDITIONS: Preterm Birth
Keywords: Pregnancy
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CenteringPregnancy group prenatal care (Experimental): Pregnant women who were randomized to receive CenteringPregnancy group prenatal care.
  Interventions: Behavioral: CenteringPregnancy
- Traditional individual prenatal care (No Intervention): Pregnant women who were randomized to receive traditional individual prenatal care.

INTERVENTIONS:
Behavioral: CenteringPregnancy — Pregnant women whose due dates are in the same month will receive ten 2-hour group prenatal care sessions according to the standard curriculum provided by the Centering Healthcare Institute.
  Arms: CenteringPregnancy group prenatal care

SUMMARY:
The purpose of the PIINC study is to identify differences in placental inflammatory lesions between women participating in group prenatal care versus standard prenatal care, and additionally, examine whether the frequency of placental inflammatory lesions differ by race and income. The investigators hypothesize that women participating in group prenatal care will have lower pro-inflammatory profiles compared to women in routine prenatal care.

DETAILED DESCRIPTION:
This is a supplementary investigation of placental inflammatory lesions among participants enrolled in a randomized controlled trial comparing biomedical, behavioral and psychosocial outcomes among pregnant women who participate in CenteringPregnancy group prenatal care, to women in the traditional individual prenatal care and to investigate whether improving women's stress, activation and engagement will explain the potential benefits of CenteringPregnancy on outcomes and health disparities. The study will be conducted in a large prenatal care center in South Carolina. Eligible White and Black women will be recruited before 20 weeks of gestational age with low risk pregnancy.

ELIGIBILITY:
Inclusion Criteria:

1. Enrollment in NICHD 1R01HD082311: Centering and Racial Disparities: A Randomized Controlled Trial on CenteringPregnancy (the "CRaDle" trial).
2. Pregnant women aged between 14-45 years
3. Enrolled in prenatal care by 20 6/7 weeks' gestation

Exclusion Criteria:

1. Medical complications of pregnancy that would preclude prenatal care provision by nurse practitioners or participation in group care

   * Pregestational diabetes,
   * Severe chronic hypertension requiring medication,
   * Morbid Obesity with BMI >49.99
   * Renal disease with baseline proteinuria >1g/24 hours
   * Any disease requiring chronic immunosuppression (SLE, solid organ transplant)
   * Active pulmonary tuberculosis
   * Sickle cell anemia
   * Human Immunodeficiency Virus Infection
   * Other medical conditions that would exclude women from group care at the discretion of the PI
2. Pregnancy complications that would preclude prenatal care provision by nurse practitioners or participation in group care

   * Multiple gestation
   * Lethal fetal anomalies
   * Other pregnancy complications that would exclude women from group care at the discretion of the PI
3. Social and behavioral complications of pregnancy which would preclude prenatal care provision by nurse practitioners or participation in group care

   * Current incarceration
   * Severe psychiatric illness

Ages: 14 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 1133 (Actual)
Dates: Start 2018-08-08 (Actual); Primary Completion 2020-10-31 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
Prevalence of placental chronic inflammatory lesions, characterized histologically | Measured at delivery
Prevalence of placental chronic inflammatory lesions stratified by placental compartment - decidua vs. villous layer vs. membranes | Measured at delivery

SECONDARY OUTCOMES:
Concentration (pg/mL) of inflammatory cytokines in peripheral maternal blood via multiplex immunoassays | Up to 43 weeks gestation
  Circulating inflammatory biomarkers C-reactive protein, IL-6, IL-8, IL-10, IL-13, INF-α, and TNF-α (pg/mL) in maternal serum will be measured during the second trimester between 20 weeks 0 days and 25 weeks and 6 days gestation, and during the third trimester between 32 weeks 0 days and 43 weeks 0 days
Differential expression of mRNA gene transcripts for 34,000 human genes | Up to 43 weeks gestation
  Characterization of transcription control differences by exposure in maternal blood via TELiS promoter sequence analysis. Pathways involved in fetal tolerance, inflammatory activity, and organ development will be characterized. Will be measured during the second trimester between 20 weeks 0 days and 25 weeks and 6 days gestation, and during the third trimester between 32 weeks 0 days and 43 weeks 0 days. The number of differentially expressed transcripts will be totaled. Differential expression will be determined by greater than or equal to a 1.25-fold differential expression between exposure groups.
Differential expression of mRNA gene transcripts for 34,000 human genes | Measured at delivery
  Characterization of transcription control differences by exposure in fresh placental biopsies via TELiS promoter sequence analysis. Pathways involved in fetal tolerance, inflammatory activity, and organ development will be characterized. The number of differentially expressed genes will be totaled. Differential expression will be determined by greater than or equal to a 1.25-fold differential expression between exposure groups.

CONTACTS AND LOCATIONS:
Overall Officials: Ann Border, MD, MSc, Principal Investigator — Endeavor Health
Locations (1):
- Greenville Health System, Greenville, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No